CLINICAL TRIAL: NCT04808882
Title: ANTIcoagulation in Severe COVID-19 Patients: a Multicenter, Parallel-group, Open-label, Randomized Controlled Trial
Brief Title: ANTIcoagulation in Severe COVID-19 Patients
Acronym: ANTICOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP201624; 2020-A03531-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2020-12

CONDITIONS: Severe COVID-19 Pneumonia
Keywords: COVID-19; Anticoagulation
MeSH Terms: conditions — COVID-19 | interventions — Tinzaparin

STUDY DESIGN:
Intervention Model Description: The research is a multicenter, parallel group, open-label, randomized controlled superiority trial, aiming at comparing three usual strategies of anticoagulation. The primary hierarchical criterion assessed at Day-28, includes all-cause mortality followed by the time to clinical improvement. The three strategies are LD-PA, HD-PA, and TA, with a 1:1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose prophylactic anticoagulation (Experimental): LD-PA
  Interventions: Drug: Tinzaparin, Low dose prophylactic anticoagulation
- High dose prophylactic anticoagulation (Experimental): HD-PA
  Interventions: Drug: Tinzaparin, High dose prophylactic anticoagulation
- Therapeutic anticoagulation (Experimental): TA
  Interventions: Drug: Tinzaparin,Therapeutic anticoagulation

INTERVENTIONS:
Drug: Tinzaparin, Low dose prophylactic anticoagulation — Participants randomized to the LD-PA strategie will receive the low weight molecular heparin (LMWH) tinzaparin, considering its contraindications, recommended dose ranges and monitoring if applicable, as follows: LD-PA : 3500 IU/24h. Depending on the type of tinzaparin pre-filled syringe available in the participating center, the dose of 4000 IU/24h will be allowed in place of 3500 IU/24h.
  If tinzaparin is not punctually available, the use of enoxaparin will be allowed as follows: LD-PA: 4000 IU/24h.
  After day-14, or hospital discharge, or in case of an indication for TA, or of serious adverse event related to anticoagulation, the investigational anticoagulation strategy will be discontinued and anticoagulation treatment will be left at the discretion of attending physicians.
  Recommendations for the management of COVID-19 pneumonia will be followed, including the use of dexamethasone. These recommendations will be subject to modifications based on the new literature data.
  Other Names: LD-PA
  Arms: Low dose prophylactic anticoagulation
Drug: Tinzaparin, High dose prophylactic anticoagulation — Participants randomized to the HD-PA strategie will receive the low weight molecular heparin (LMWH) tinzaparin, considering its contraindications, recommended dose ranges and monitoring if applicable, as follows: HD-PA : 7000 IU/24h.
  If tinzaparin is not punctually available, the use of enoxaparin will be allowed as follows: HD-PA: 4000 IU/12h.
  After day-14, or hospital discharge, or in case of an indication for TA, or of serious adverse event related to anticoagulation, the investigational anticoagulation strategy will be discontinued and anticoagulation treatment will be left at the discretion of attending physicians.
  Recommendations for the management of COVID-19 pneumonia will be followed, including the use of dexamethasone. These recommendations will be subject to modifications based on the new literature data.
  Other Names: HD-PA
  Arms: High dose prophylactic anticoagulation
Drug: Tinzaparin,Therapeutic anticoagulation — Participants randomized to the TA strategie will receive the low weight molecular heparin (LMWH) tinzaparin, considering its contraindications, recommended dose ranges and monitoring if applicable, as follows: TA : 175 IU/kg/24h.
  If tinzaparin is not punctually available, the use of enoxaparin will be allowed as follows: TA: 100 IU/kg/12h.
  After day-14, or hospital discharge, or in case of an indication for TA, or of serious adverse event related to anticoagulation, the investigational anticoagulation strategy will be discontinued and anticoagulation treatment will be left at the discretion of attending physicians.
  Recommendations for the management of COVID-19 pneumonia will be followed, including the use of dexamethasone. These recommendations will be subject to modifications based on the new literature data.
  Other Names: TA
  Arms: Therapeutic anticoagulation

SUMMARY:
Coronavirus disease 2019 (COVID-19), a viral respiratory illness caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), may predispose patients to thrombotic disease due to a state of profound inflammation, platelet activation, and endothelial dysfunction leading to respiratory distress and increased mortality. The incidence of macrovascular thrombotic events varies from 10 to 30% in COVID-19 hospitalized patients depending on the type of arterial or vein thrombosis captured and severity of illness . Observational results in patients receiving routine low-dose prophylactic anticoagulation (LD-PA), several institutions have recently released guidance statement to prevent macrovascular thrombotic events with dose escalation anticoagulation. In these recommendations, high-dose prophylactic anticoagulation (HD-PA) and therapeutic anticoagulation (TA) can be employed either empirically or based on the body mass index and increased D-dimer values. No randomized trial has validated this approach, and other recent recommendations challenge this approach. Microvascular thrombotic events are also of major concern in critically ill patients with COVID-19, even in the absence of obvious macrovascular thrombotic events. A large review of autopsy findings in COVID-19-related deaths reported micro thrombi in small pulmonary vessels. More generally, COVID-19-induced endothelitis and coagulopathy across vascular beds of different organs lead to widespread microvascular thrombosis with microangiopathy and occlusion of capillaries. Thus, in severe COVID-19 patients requiring oxygen therapy without initial macrovascular thrombotic event, a HD-PA or a TA could be beneficial by limiting the extension of microvascular thrombosis and the evolution of the lung and multi-organ microcirculatory dysfunction. In a large observational cohort of 2,773 COVID-19 patients, a lower in-hospital mortality in ventilated patients receiving TA as compared to those receiving PA (29.1% vs. 62.7%). Our hypothesis is dual: i) first, that TA and HD-PA strategies mitigate microthrombosis and each limit the progression of COVID-19, including respiratory failure and multi-organ dysfunction, with in fine a decreased mortality and duration of disease, as compared to a low-dose PA; ii) second, that TA outperforms HD-PA in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* Severe COVID-19 pneumonia, defined by:

  * A newly-appeared pulmonary parenchymal infiltrate; AND
  * a positive RT-PCR (either upper or lower respiratory tract) for COVID-19 (SARS-CoV-2); AND
  * WHO progression scale ≥ 5 (on The Who ordinal scale)
* Written informed consent (patient, next of skin or emergency situation).
* In view of the exceptional and urgent situation, affiliation to a social security scheme will not be a criterion for inclusion.

Exclusion Criteria:

* Pregnancy and breast feeding woman;
* Postpartum (6 weeks);
* Extreme weights (<40 kg or >100 kg);
* Patients admitted since more than 72 hours to the hospital (if the WHO ordinal scale is 5 at time of inclusion) or since more than 72 hours to the intensive care unit (if the WHO ordinal scale is 6 or more at time of inclusion);
* Need for therapeutic anticoagulation (except for COVID-related pulmonary thrombosis);
* Bleeding event related to hemostasis disorders, acute clinically significant bleed, current gastrointestinal ulcer or any organic lesion with high risk for bleeding
* Platelet count < 50 G/L;
* Within 15 days of recent surgery, within 24 hours of spinal or epidural anesthesia;
* Any prior intracranial hemorrhage, enlarged acute ischemic stroke, known intracranial malformation or neoplasm, acute infectious endocarditis;
* Severe renal failure (creatinine clearance <30 mL/min);
* Iodine allergy;
* Hypersensitivity to heparin or its derivatives including low-molecular-weight heparin;
* History of type II heparin-induced thrombocytopenia;
* Chronic oxygen supplementation;
* Moribund patient or death expected from underlying disease during the current admission;
* Patient deprived of liberty and persons subject to institutional psychiatric care;
* Patients under guardianship or curatorship;
* Participation to another interventional research on anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Day-28
Number of days to clinical improvement | Day-28
  Clinical improvement will be assessed through a seven-category ordinal scale derived from the WHO scale, using the following categories: 1. not hospitalized with resumption of normal activities; 2. not hospitalized, but unable to resume normal activities; 3. hospitalized, not requiring supplemental oxygen; 4. hospitalized, requiring supplemental oxygen; 5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6. hospitalized, requiring ECMO, invasive mechanical ventilation, or both; and 7. death. As all included patients will at least require oxygen supplementation, live discharge from hospital will represent a minimal 2-points decrease in the 7-points scale, thus a clinical improvement.

SECONDARY OUTCOMES:
Net clinical benefit of anticoagulation assessed by the absence of thrombotic event, major bleeding event, Heparin Induced Thrombocytopenia and all-cause death | Day-28
All-cause deaths | Day-28 and Day-90
Proportion of patients with at least one thrombotic event at Day-28 | Day-28
Proportion of patients with at least one major bleeding event (MBE) at Day-28 | Day-28
Proportion of patients with at least one life-threatening bleeding event at Day-28 | Day-28
Proportion of patients with any bleeding event at Day-28 | Day-28
Proportion of patients with Heparin Induced Thrombocytopenia at Day-28 | Day-28
Number of days to clinical improvement assessed through a seven-category ordinal scale derived from the WHO scale | Day-28
Score on the seven-category ordinal scale derived from the WHO Ordinal scale | Day-28
Score on WHO Ordinal Scale | Day-28
Number of days alive and free from supplemental oxygen at Day-28 | Day-28
Proportion of patients needing intubation at Day-28 | Day-28
Number of days alive and free from invasive mechanical ventilation at Day-28 | Day-28
Number of days alive and free from vasopressors at Day-28 | Day-28
Length of intensive care unit stay | Day-28
Length of hospital stay | Day-28
Quality of life and disability at assessed using a quality of life questionnaire | Day-90
D-dimers levels | Day-7
Sepsis-Induced Coagulopathy Score (SCS) | Day-7

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LABBE, MD, Study Director — Assistance Publique Hopitaux de Paris (AP-HP)
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] Labbe V, Contou D, Heming N, Megarbane B, Razazi K, Boissier F, Ait-Oufella H, Turpin M, Carreira S, Robert A, Monchi M, Souweine B, Preau S, Doyen D, Vivier E, Zucman N, Dres M, Fejjal M, Noel-Savina E, Bachir M, Jaffal K, Timsit JF, Picos SA, Mariotte E, Martis N, Juguet W, Melica G, Rondeau P, Audureau E, Mekontso Dessap A; ANTICOVID Investigators. Effects of Standard-Dose Prophylactic, High-Dose Prophylactic, and Therapeutic Anticoagulation in Patients With Hypoxemic COVID-19 Pneumonia: The ANTICOVID Randomized Clinical Trial. JAMA Intern Med. 2023 Jun 1;183(6):520-531. doi: 10.1001/jamainternmed.2023.0456. PMID 36946232
- [Derived] Labbe V, Contou D, Heming N, Megarbane B, Ait-Oufella H, Boissier F, Carreira S, Robert A, Vivier E, Fejjal M, Doyen D, Monchi M, Preau S, Noel-Savina E, Souweine B, Zucman N, Picos SA, Dres M, Juguet W, Mariotte E, Timsit JF, Turpin M, Razazi K, Gendreau S, Baloul S, Voiriot G, Fartoukh M, Audureau E, Mekontso Dessap A. Comparison of standard prophylactic, intermediate prophylactic and therapeutic anticoagulation in patients with severe COVID-19: protocol for the ANTICOVID multicentre, parallel-group, open-label, randomised controlled trial. BMJ Open. 2022 Apr 26;12(4):e059383. doi: 10.1136/bmjopen-2021-059383. PMID 35473740